CLINICAL TRIAL: NCT02126176
Title: Protopic Adherence and Efficacy in Korean Eczema Patient
Status: Completed | Type: Observational
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUNHDM-adherence
Record Dates: First submitted 2014-04-24; First posted 2014-04-29 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether the dosage of 0.1% tacrolimus ointment applied on unit area of eczema influence the efficacy of treatment.

ELIGIBILITY:
Inclusion Criteria:

* at least 19 years of age with a diagnosis of atopic dermatitis
* treated with protopic 0.1% ointment

Exclusion Criteria:

* treated with other medication or topical agent
* skin lesion on the scalp or hand and foot
* pregnant women/lactating women

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with atopic dermatitis
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
clinical assessments of erythema, scaling, and pruritus | 2 weeks
  EASI score
clinical assessments of erythema, scaling, and pruritus | 2 weeks
  TIS score
clinical assessments of erythema, scaling, and pruritus | 2 weeks
  IGA/PGA score
clinical assessments of erythema, scaling, and pruritus | 2 weeks
  DLQI
clinical assessments of erythema, scaling, and pruritus | 2 weeks
  itching VAS scale

CONTACTS AND LOCATIONS:
Locations (1):
- Department of dermatology, Pusan National University Hospital, Busan, Busan, South Korea